CLINICAL TRIAL: NCT05539222
Title: The Effect of Food Vouchers and an Educational Intervention on Promoting Healthy Eating in Vulnerable Groups. A Pilot Study
Brief Title: Food Vouchers and Educational Intervention on Promoting Healthy Eating in Vulnerable Groups.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, María Isabel Iguacel Azorín, Associate Professor, Universidad de Zaragoza
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: PI20/541
Record Dates: First submitted 2022-09-01; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Economic Problems
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food voucher plus health and nutritional education (Active Comparator): Intervention and control group individuals received 120 euros/month during 3 months in food vouchers to be spent in supermarkets (60 euros/month if under 12y) plus a 10-week nutrition education for the intervention group.
  Interventions: Other: Food vouchers and education
- Food voucher (No Intervention): Intervention and control group individuals received 120 euros/month during 3 months in food vouchers to be spent in supermarkets (60 euros/month if under 12y) plus a 10-week nutrition education for the intervention group.

INTERVENTIONS:
Other: Food vouchers and education — Intervention and control group individuals received 120 euros/month during 3 months in food vouchers to be spent in supermarkets (60 euros/month if under 12y) plus a 10-week nutrition education for the intervention group. Family food purchases were assessed using electronically recorded supermarket-obtained transactions.
  Arms: Food voucher plus health and nutritional education

SUMMARY:
Cost has been reported as the main barrier to healthy eating in vulnerable groups. We aimed to evaluate the effect of food vouchers with a nutrition education intervention on diet quality (using NOVA classification) and health. This pilot study has a randomized pre-and post-test experimental design. We included 66 vulnerable users from the Red Cross of Zaragoza (Spain). Intervention and control group individuals received 120 eu-ros/month during 3 months in food vouchers to be spent in supermarkets (60 eu-ros/month if under 12y) plus a 10-week nutrition education for the intervention group. Family food purchases were assessed using electronically recorded supermarket-obtained transactions. We found the percentage of healthy food was higher in the in-tervention group than in the control group. Once the nutrition education was over, dif-ferences between groups dissipated. Health parameters improved in the intervention group, particularly weight-status, lipid, and liver enzymes. Control participants gained weight, although lipid and liver enzymes improved. Blood pressure and HbA1c did not improve in either the intervention or the control group. In conclusion, providing unrestricted food vouchers to vulnerable groups to increase healthy food consumption and reduce the intake of ultra-processed food appears to be insufficient and should be accompanied by medium-long term education.

ELIGIBILITY:
Inclusion Criteria: The inclusion criteria established were children and adults between 3 and 80 years of age with at least one adult per family unit that could speak and understand Spanish, French, or English.

Exclusion Criteria: Adults with severe illness or cognitive impairment were excluded from the study.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Diet quality (using NOVA classification) | 3 months
  For the analysis of the products purchased by the family unit, the NOVA food classification was used. This classification groups products according to their degree of manufacture so that Group 1 are those products that are unprocessed or minimally processed; Group 2 are culinary processed products or food industry ingredients (oil, sugar, honey, salt, butter); Group 3 are products processed from Group 1 foods, such as canned vegetables, nuts with salt or fish preserved in oil or water; and Group 4 are ultra-processed products [23]. The rationale and details on each NOVA food group have been described elsewhere [24]. Two investigators classified each food item according to the NOVA classification criteria, and for some items with discrepant classification, they were resolved by discussion. Non-food items (e.g. cleaning products and other products that were purchased with the non-food voucher) were classified as "Others".
Adherence Mediterranean diet | 10-week
  To determine the degree of adherence to the Mediterranean diet, a specific short questionnaire of fourteen items validated for the Spanish population and used by the Prevention with Mediterranean Diet (PREDIMED) group was used. To obtain the score, a value of +1 is assigned to each of the items with a positive connotation with re-spect to DM and -1 when the items have a negative connotation. In adults, from the sum of the values obtained in the 14 items, the degree of adherence is determined, establishing two levels, so that if the total score is greater than or equal to nine, it is a diet with a good level of adherence, and if the total sum is less than nine, the diet has a low level of adherence.
  In children, the questionnaire consist of 16 questions and two possible answer options (yes/no), with 12 positive and 4 negative questions.
  The levels of adherence to the Mediterranean diet were classified into three groups: poor (0-3), average (4-7) and good (8-12).

SECONDARY OUTCOMES:
Weight | 10-week
  Anthropometric data included body weight and height presented to the nearest 0.01 kg and 0.01 mm, respectively. Body Mass Index (BMI) was also calculated as body weight in kilograms divided by body height in meters squared (kg/m2). and categorized into underweight (if BMI<18.5), normal weight (18.5-24.9), overweight (25-29.9) and obesity (30 or greater). BMI for children and adolescents was converted to an age- and sex-specific z-score using the extended IOTF criteria. To assess weight and body composition, the TANITA MC780SMA portable beam scale was used.
Height | 10-week
  Anthropometric data included body weight and height presented to the nearest 0.01 kg and 0.01 mm, respectively. Body Mass Index (BMI) was also calculated as body weight in kilograms divided by body height in meters squared (kg/m2). and categorized into underweight (if BMI<18.5), normal weight (18.5-24.9), overweight (25-29.9) and obesity (30 or greater). BMI for children and adolescents was converted to an age- and sex-specific z-score using the extended IOTF criteria. To assess weight and body composition, the TANITA MC780SMA portable beam scale was used.
Blood pressure | 10-week
  Systolic blood pressure (SBP) and diastolic blood pressure (DBP) in mmHg were measured with an automatic oscillometric device (OMRON M6). All participants were asked to sit for at least 5 min before taken the measurement. Two measurements were taken with a 2-minute interval plus a further measurement in case of a >5% difference in blood pressure between the first two readings. The average of the two (or three) measurements was used for statistical analysis.
Uric acid | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
Blood urea nitrogen (BUN) | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
ALP (Alkaline phosphatase) | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
ALT (alanine transaminase) | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
AST (aspartate aminotransferase) | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
Gamma-glutamyl transferase (GGT) | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
Triglycerides | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
Total cholesterol (TC) | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
High-density lipoprotein cholesterol (HDL-C) | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
Low-density lipoprotein cholesterol (LDL-C)), | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
Fasting glucose | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.
Glycated hemoglobin A1c (HbA1c) | 10-week
  Blood samples were taken by a hematologist after 8 hours of fasting. Blood sam-ples were obtained at 9 am at pre- and post-intervention. Further, all participants were required to fast for 8 hours before extracting their blood sample. Approximately 10 mL of blood was extracted from the median antecubital vein and stored in an EDTA tube. The plasma was centrifuged for 15 minutes at 3,000 rpm at 4°C. Thereafter, the samples were stored frozen for subsequent analysis. All samples were measured directly by an automatic hematology analyzer. The laboratory carries out quality control according to standard procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- María Isabel Iguacel Azorín, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol